CLINICAL TRIAL: NCT03370367
Title: Double Blind Phase III Trial of Effects of Low Dose 13-Cisretinoic Acid on Prevention of Second Primaries in Stages I-II Head and Neck Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: C0590
Record Dates: First submitted 2017-12-07; First posted 2017-12-12 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Stage I-II Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Isotretinoin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A (Experimental): 13-cis retinoic acid will be dispensed in 3.75 mg and 5 mg gelatin capsules. Take 2 capsules once a day for up to 2 years.
  Interventions: Drug: 13-cis retinoic acid
- Arm B (Placebo Comparator): Take 2 placebo pills once a day for up to 2 years.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: 13-cis retinoic acid — Taken daily.
  Arms: Arm A
Other: Placebo — Placebo
  Arms: Arm B

SUMMARY:
In this trial the investigators propose to utilize 13-cRA to prevent dysplastic changes and second malignancies in patients with squamous cell carcinoma of the head and neck regions who have a high probability of cure from their primary cancer. Comparisons between patients treated by 13-cRA and patients receiving placebo will include:

1. The time to diagnosis of second primary for the treatment versus control groups.
2. Survival time for the treatment versus control groups.
3. Secondarily, the cost-benefit ratio for 13-cRA will be analyzed by assessing the toxicities of 13-cis retinoic acid treated patients in comparison to those experienced by placebo treated patients.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent i obtained, the approved form is signed, and on file at the institution.
* Histologically confirmed squamous cell carcinoma.
* All chest x-rays and cervical spine x-rays done after definitive treatment within 35 days prior to randomization and all hematology andchemistries done within 2 weeks prior to randomization.
* The following sites and stages of cancers will be eligible. Oral Cavity

  1. T1 NO
  2. T2 NO 3.142 Oropharynx

  <!-- -->

  1. T1 NO
  2. T2 NO 3.143 Hypopharynx

  1. T1 NO 3.144 Larynx
  1. T1 NO
  2. T2 NO
* Age greater than 18 years.
* ECOG performance status 0 or 1.
* Patients must have adequate bone marrow, hepatic and renal function defined as follows: WBC >3,500/mm, Platelets > 125,000/mm.3 Total Bilirubin < 2 mg%, Serum creatinine < 2.5 mg%. Serum SGOT < 2x normal, Alkaline Phosphatase < 2x normal. Fasting Serum triglyceride levels < 210 mg %. Fasting cholesterol < 350 mg %. Patient may not be under systemic therapy for hyperlipidemia or have symptomatic arteriosclerotic coronary artery disease or have undergone coronary bypass surgery.
* The patient must have completed primary treatment of their cancer with surgery and/or radiation therapy within 730 days prior to randomization.
* The patient has had surgery and/or radiation therapy as outlined in Sections 5.0 and 6.0, and has been rendered disease-free.
* If currently receiving, patient must discontinue mega vitamin doses

Exclusion Criteria:

* Women of child bearing potential.
* Patient with severe coronary artery disease (Class III-IV New York Heart Association.)
* Histology other than squamous cell carcinoma.
* Distant metastases.
* Completion of previous treatment for their primary cancer with radiation, or surgery (except for biopsy) more than 730 days ago.
* Prior, synchronous, or concurrent malignancy except basal cell skin cancer.
* Failure to be rendered disease-free of primary tumor (includes positive surgical margins).
* The patient has had prior therapy other than that outlined in Sections 5.0 and 6.0 of the protocol.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 1989-05-15 (Actual); Primary Completion 1999-01-15 (Actual); Study Completion 2015-04-14 (Actual)

PRIMARY OUTCOMES:
The time to diagnosis of second primary for the treatment versus control groups. | 20 years

SECONDARY OUTCOMES:
Survival time for the treatment versus control groups. | 20 years

REFERENCES:
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/